CLINICAL TRIAL: NCT06305585
Title: Can a Manual Therapy Technique Help Relieve Stress? Assessing Effects of Primal Reflex Release on the Body's Stress Response
Brief Title: Can a Novel Manual Therapy Technique Help Relieve Stress? Assessing Effects of Primal Reflex Release on the Body's Stress Response
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Idaho (Other)
Collaborators: CJ Brush (Unknown); Jayme Baker (Unknown); Sydney Leverett (Unknown)
Responsible Party: Principal Investigator, Nickolai Martonick, Assistant Professor, University of Idaho
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB# 23-214
Record Dates: First submitted 2024-02-28; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Psychological Stress
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primal Reflex Release Technique (Experimental): The subject will lay on their back with their eyes closed. Palmar Reflex Release The subject will actively raise arms overhead (palm facing the floor) with a pen squeezed between their fingers.
  Epicranial Release The clinician will grasp the subject's hair near the front of the hairline with one hand, just above the ear on the right side and gently pull.
  Frontalis Release The clinician will instruct the subject to raise their eyebrows and keep them raised. The clinician will use their thumbs to gently flick downward on the inside portion of the subject's eyebrows.
  Orbicularis Oculi Release The clinician will place their thumb below the eye resting on the cheek bone and with the other hand will lightly rest on the subject's eyelid The clinician will then gently and lightly attempt to quickly open the subject's eyelids
  Suboccipital Release The participant will rest their head in clinicians hands while they provide a slight traction at the base of the skull
  Interventions: Other: Primal Reflex Release Technique (PRRT)
- Control (No Intervention): For the control, the subject will watch another 5-minute video of fish in an aquarium.

INTERVENTIONS:
Other: Primal Reflex Release Technique (PRRT) — Primal Reflex Release Technique (PRRT) is a non-invasive complementary hands-on treatment method intended to help relax the central nervous system by gently stimulating innate protective reflexes. A certified practitioner applies light tactile stimulation to targeted areas in a structured sequence postulated to help release hypertonic muscles, restore regulation of automatic responses, and enable a calm, parasympathetic state.
  Arms: Primal Reflex Release Technique

SUMMARY:
Stress, when left unmanaged, can have detrimental effects on both physical and mental health, contributing to conditions such as high blood pressure, anxiety, and even cardiovascular disease. Effective stress management therapies may help maintain overall well-being and reduce the risk of long-term health complications. The Primal Reflex Release Technique (PRRT) is a novel manual therapy that may reduce markers related to stress such as heart rate variability (HRV) and patient-reported outcomes (PROs). Therefore, the purpose of this study is to elucidate the potential for PRRT to improve HRV and PROs.

DETAILED DESCRIPTION:
This randomized, controlled experimental intervention study evaluates acute impacts of a reflex-targeted manual therapy called Primal Reflex Release Technique (PRRT) on cardiovascular indices of stress and sympathetic tone. After consenting and baseline characteristics, subjects are allocated to receive either the PRRT or the control condition.

Continuous electrocardiography (ECG) and impedance cardiography (ICG) monitoring will be used to track heart rate variability (HRV) changes across three phases:

1. Pre-intervention during a 5-minute video of aquatic nature scenes to establish resting baseline
2. 5 minutes of a practitioner administering targeted spinal manipulation PRRT protocol in the treatment group to stimulate innate protective reflexes OR continued relaxation video viewing for control group
3. Post-intervention repeat of the standardized video to assess changes after PRRT session without ongoing manipulation

The PRRT targets precise anatomical locations and neural pathways including stimulating facial muscles, upper spinal reflexes and traction of the suboccipital muscles. Brief, reversible sensations will occur without expected harm or lasting effects.

Psychological state assessed via paper mood scales pre/post tracks subjective stress correlates. Analysis using linear mixed effects models contrast whether indices of cardiovascular reactivity and psychological responses shift acutely with PRRT versus control video. Findings could provide physiological validation for integration as stress-alleviating treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject can refrain from caffeinated beverages in the 6 hours prior to data collection
* Subject is not currently taking any beta blockers
* Subject is comfortable with a manual therapy technique where the clinician touches your face and head

Exclusion Criteria:

* Subject has had caffeine within 6 hours
* Subject is currently taking any beta blockers

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
ECG Data | Through study completion, an average of 6 months.
  ECG will be used to derive respiratory sinus arrythmia (RSA), which will be derived as the natural-logged spectral power value in the high-frequency bandwidth (0.15-0.40 Hz).
ICG Data | Through study completion, an average of 6 months.
  ICG will be used to derive pre-ejection period (PEP), which represents the time between the onset of ventricular depolarization and the opening of the aortic valve.
Depression Anxiety Stress Scale-21 (DASS-21) - Depression | Through study completion, an average of 6 months.
  The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress. Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content. The depression scale assesses dysphoria, hopelessness, devaluation of life, self-deprecation, lack of interest / involvement, anhedonia and inertia. Scores for depression are calculated by summing the scores for the relevant items (0-42) with higher scores indicating greater levels of depression.
Depression Anxiety Stress Scale-21 (DASS-21) - Anxiety | Through study completion, an average of 6 months.
  The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress. Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content. The anxiety scale assesses autonomic arousal, skeletal muscle effects, situational anxiety, and subjective experience of anxious affect. Scores for anxiety are calculated by summing the scores for the relevant items (0-42) with higher scores indicating greater levels of anxiety.
Depression Anxiety Stress Scale-21 (DASS-21) - Stress | Through study completion, an average of 6 months.
  The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress. Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content. The anxiety scale assesses autonomic arousal, skeletal muscle effects, situational anxiety, and subjective experience of anxious affect. The stress scale is sensitive to levels of chronic nonspecific arousal. It assesses difficulty relaxing, nervous arousal, and being easily upset / agitated, irritable / over-reactive and impatient. Scores for stress are calculated by summing the scores for the relevant items (0-42) with higher scores indicating greater stress.
Simple Physical Activity Questionnaire (SIMPAQ) | Through study completion, an average of 6 months.
  The SIMPAQ is used to determine the average amount of time that participants spend exercising per day.
Self Assessment Manikin (SAM) - Valence | Through study completion, an average of 6 months.
  Assessment of valence ranging on a 9-point scale from 1 (feeling pleasant) to 9 (feeling unpleasant).
Self Assessment Manikin (SAM) - Arousal | Through study completion, an average of 6 months.
  Assessment of arousal ranging on a 9-point scale from 1 (feeling excited) to 9 (feeling calm).

CONTACTS AND LOCATIONS:
Locations (1):
- ISMaRT Clinic, Moscow, Idaho, United States

IPD SHARING:
Plan to Share IPD: No